CLINICAL TRIAL: NCT02398084
Title: Particle Sizing of Masticated Tree Nuts - Cashews and Walnuts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14/LO/2286
Record Dates: First submitted 2015-03-11; First posted 2015-03-25 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: mastication; cashews; walnuts; participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chewing of nuts (Experimental): 8 samples (4-5 g) of nuts (cashews or walnuts) on two separate visit days.
  Interventions: Other: Chewing of nuts

INTERVENTIONS:
Other: Chewing of nuts — The volunteers will be asked to chew and spit 8 portions (4-5 g) of nuts (cashews or walnuts) on two separate visits. They will provide samples for particle sizing. Two portions will be used as practice samples in order to measure the number of chews. Two portions will be sieved. Two portions will be measured by laser diffraction. Two portions will be frozen for later lipid analysis.

SUMMARY:
The investigators want to understand how oral processing (chewing) of nuts affects particle size and the presence of lipid (fat) on the cut surfaces.

The main objective of the study is to:

Measure the size of nut particles that have been chewed sufficiently to be swallowed.

The secondary objective of this study is to:

Measure any changes in lipid content due to chewing and compare it to a prediction from a theoretical model.

The investigators have developed a theoretical model for determining the release of nutrients from plant foods, specifically lipid (fat) from almonds. The model has been used to calculate the amount of lipid released from chewed almonds. The model shows that only about 10% of the lipid is immediately released. The investigators require information on the particle size distribution (number of particles of each size) for other chewed nuts to calculate the amount of lipid released for other nuts. This will allow us to check the validity of our model for other foods.

ELIGIBILITY:
Inclusion Criteria:

* Must be generally healthy
* Must have eaten nuts within the last month with no adverse effects

Exclusion Criteria:

* Must not be allergic to nuts of any kind
* Must not have any teeth missing (apart from unerupted wisdom teeth)
* Must not have bleeding gums
* Must not have had dental treatment (other than checkups) in the last 3 months
* Must not be currently suffering from any infectious disease that may be passed on via saliva e.g. Glandular fever, flu

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Particle size distribution of masticated nuts | At time of expectoration, up to 90 seconds after each sample ingested.
  Particle size distribution of masticated nuts as measured by laser diffraction and sieving.

SECONDARY OUTCOMES:
Lipid content of masticated nuts | At time of expectoration, up to 90 seconds after each sample ingested.
  Lipid content of masticated nuts as measured by Soxhlet to be compared to predictions form mathematical model.

CONTACTS AND LOCATIONS:
Overall Officials: Terri Grassby, BSc PhD, Principal Investigator — King's College London
Locations (1):
- Diabetes and Nutritional Sciences Division, School of Medicine, King's College London, London, United Kingdom

REFERENCES:
- [Background] Grundy MM, Grassby T, Mandalari G, Waldron KW, Butterworth PJ, Berry SE, Ellis PR. Effect of mastication on lipid bioaccessibility of almonds in a randomized human study and its implications for digestion kinetics, metabolizable energy, and postprandial lipemia. Am J Clin Nutr. 2015 Jan;101(1):25-33. doi: 10.3945/ajcn.114.088328. Epub 2014 Nov 12. PMID 25527747
- [Background] Grassby T, Picout DR, Mandalari G, Faulks RM, Kendall CW, Rich GT, Wickham MS, Lapsley K, Ellis PR. Modelling of nutrient bioaccessibility in almond seeds based on the fracture properties of their cell walls. Food Funct. 2014 Dec;5(12):3096-106. doi: 10.1039/c4fo00659c. PMID 25310222